CLINICAL TRIAL: NCT00205413
Title: Low Dose Helical Computed Tomographic (CT) Screening Followed by Anatomic Co-Registered Computed Tomography With Positron Emission Tomography (CT/PET) for Patients With Indeterminate (5-9 mm) Nodules
Brief Title: Surveillance For New Lung Primaries
Status: Terminated | Type: Observational
Why Stopped: low accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2002-376
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Lung Cancer
Keywords: surveillance for lung cancer
MeSH Terms: conditions — Lung Neoplasms

SUMMARY:
This clinical research protocol proposes to perform low dose helical computed tomographic (CT) scanning in 250 high-risk patients (125/year for two years) in order to detect lung carcinomas when they are small and subject to effective curative therapies.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic

Exclusion Criteria:

* 20 pack year history

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2002-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Weigel, MD, Principal Investigator — University of Wisconsin Medical School
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States